CLINICAL TRIAL: NCT07205770
Title: Comparison of Proprioceptive Neuromuscular Facilitation and Passive Stretching Methods in Individuals With Scoliosis
Brief Title: Comparison of Stretching Methods in Individuals With Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gönül Elpeze (Other)
Responsible Party: Sponsor-Investigator, Gönül Elpeze, Assistant Proffessor, Gaziantep Islam Science and Technology University
Organization: Gaziantep Islam Science and Technology University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Scoliosis
Record Dates: First submitted 2025-09-11; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis Idiopathic Adolescent Treatment
Keywords: scoliosis; flexibility; stretching; PNF
MeSH Terms: conditions — Scoliosis | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Stretching
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proprioceptif Neuromuscular Facilitation Stretching (Experimental): Applying 30 seconds
  Interventions: Other: PNF
- Passive Stretching Exercise (Active Comparator): Applying 30 seconds
  Interventions: Other: Passive Stretching

INTERVENTIONS:
Other: PNF — Applying to the extensor muscles for 30 seconds
  Arms: Proprioceptif Neuromuscular Facilitation Stretching
Other: Passive Stretching — Applying to the extensor muscles for 30 seconds
  Arms: Passive Stretching Exercise

SUMMARY:
The goal of this research study is to learn about the comparison of Stretching Methods in individuals with scoliosis aged of 14-65, who receive intervention Proprioceptive Neuromuscular Facilitation and Passive Stretching. The main question it aims to answer is:

Does ankle exercise lower knee joint proprioception and pain in individuals with knee pain? Does intervention Proprioceptive Neuromuscular Facilitation affect the position of the head, endurance of the spine in individuals with scoliosis? Researchers will compare Proprioceptive Neuromuscular Facilitation (the intervention) with Passive Stretching (as part of their regular medical care for scoliosis) to determine if Proprioceptive Neuromuscular Facilitation is effective in improving the position of the head, endurance of the spine.

Participants will be asked to do exercises and to let the researchers to take their measurements.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Having been diagnosed with scoliosis
* Having a Cobb angle ≤ 10°

Exclusion Criteria:

* Having undergone scoliosis surgery
* Having structural scoliosis
* Having used a brace in the last 6 months or currently using one.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
flexibility of the spine | Baseline and 6 weeks
  Modify Schobber Test
The position of the head | Baseline and 6 weeks
  Tragus-wall distance

SECONDARY OUTCOMES:
Endurance of the spine | Baseline and 6 weeks
  Biering-Sorenson Test
Cervical ROM | Baseline and 6 weeks
  Universal gonyometer

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Islam Science and Technology University, Gaziantep, Turkey (Türkiye)